CLINICAL TRIAL: NCT01483209
Title: Treatment of Vasopressor-induced Ischemia With Botulinum Toxin A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032002
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Ischemia; Vasopressor
Keywords: Digital ischemia; Vasopressor
MeSH Terms: conditions — Ischemia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botox injection (Experimental): Use of botulinum toxin A to determine efficacy in treating vasopressor-induced digital ischemia
  Interventions: Drug: Injection of botulinum toxin A

INTERVENTIONS:
Drug: Injection of botulinum toxin A — One-time injection of 100 units of botulinum toxin into hand to perform full chemical digital sympathectomy
  Other Names: Botox

SUMMARY:
The goal of this project is to determine if performing a "chemical sympathectomy" by injecting botulinum toxin A in critically ill patients on vasopressors can treat digital ischemia. This is a prospective, non-randomized pilot study designed to demonstrate proof of concept. We propose to study patients in the intensive care units of Duke Hospital who, secondary to exposure to vasoactive medications used to maintain acceptable blood pressures, have developed signs and symptoms of digital ischemia. A paired T-test will be used to compare pre- and post-injection Laser Doppler measurements for the experimental hand. We will again use a paired t-test to compare the experimental hand against the contralateral control hand. There were no major adverse events reported by the product information sheet or in other related studies of Botox for digital ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted to the ICU
* Have digital ischemia and
* Be on a vasopressor infusion

Exclusion Criteria:

* Patients with a history of systemic sclerosis
* Patients actively receiving aminoglycoside antibiotics - aminoglycosides may potentiate the effect of Botox
* Patients who have previously received botulinum toxin (A or B) injections
* Patients with a history of disorders of neuromuscular transmission (e.g myasthenia gravis, Lambert-Eaton, etc.) - Botox may have a lasting effect in these patients given their disorder
* Patients with clinical evidence of an infection in either forearm or hand
* Patients with a history of sensitivity to albumin - Botox is sold in powder form and there is albumin in the formulation
* Pregnancy - Botox is a class C medication
* Rheumatoid Arthritis
* Upper extremity arterio-venous graft or fistula
* Digital necrosis
* History of hand amputation
* Patients whom the intensive care attending physician deems will expire within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Shortell, MD, Principal Investigator — Duke UMC; Detlev Erdmann, M.D., Ph. D., Study Director — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Boxtox Injection: Subjects will serve as their own controls. Both hands are evaluated and the hand demonstrating more severe ischemia will be the one to receive the Botox (experimental treatment).
Period: Overall Study
Arm/Group | Boxtox Injection
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Boxtox Injection
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Perfusion (as Determined by Laser Doppler Measurements)
Description: A paired T-test will be used to compare pre- and post-injection Laser Doppler measurements for the experimental hand. We will again use a paired t-test to compare the experimental hand against the contralateral control hand. Results for the experimental and control groups will be plotted and displayed graphically as percent change in Doppler flow (y-axis) and time (x-axis).
Time Frame: 12 months
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Botox Injection
Number analyzed (Participants) | 0

2. Secondary Outcome: Digital Amputations
Description: The number of digits amputated in our patient cohort is a secondary endpoint of this study. We will use a paired t-test to compare the number of digital amputations in the control versus experimental group.
Time Frame: 12 months
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Botox Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Botox Injection
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Due to low accrual for this study we were unable to perform any data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes